CLINICAL TRIAL: NCT06491784
Title: EXercise TheRApy in Mesothelioma - A Feasibility Study
Brief Title: EXTRA-Meso (EXercise TheRApy in Mesothelioma) Feasibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Surrey (Other); Manchester University NHS Foundation Trust (Other Government); Mesothelioma UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GN22ON168
Record Dates: First submitted 2024-03-27; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: 1:1 randomisation, feasibility study
Masking Description: Open label, no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Routine clinical follow-up
- Exercise Therapy (Intervention) (Active Comparator): 12 week multi-modal exercise and wellbeing programme
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Other: Exercise Therapy — 12 week personalised exercise, nutrition and wellbeing programme
  Arms: Exercise Therapy (Intervention)

SUMMARY:
The goal of this clinical trial is to learn whether running an exercise study in patients with mesothelioma is feasible. The main question(s) it aims to answer are:

1. Is it feasible to recruit patients to a randomised clinical trial of exercise therapy
2. What are the barriers to study recruitment
3. What are the barriers to study retention

Participants who decide to take part in the study will be randomly allocated one of two study arms:

1. Standard of care, where the participant will undergo their usual clinical follow-up
2. Exercise therapy, where the participant will receive a personalised 12 week exercise, nutrition and wellbeing programme Participants in both study arms will be asked to complete quality of life questionnaires and a basic fitness assessment at the start and end of the study follow-up period.

Participants will be asked if they would be happy to conduct a short interview with a member of the research team, to assess their views on the study. This interview will be audio recorded and the audio recording will be transcribed anonymously to allow researchers to improve future study design.

DETAILED DESCRIPTION:
The aim of this study is to examine the feasibility of a randomised trial of exercise therapy in Mesothelioma. It will define likely rate of recruitment based on performance in two mesothelioma centres and identify barriers to recruitment and retention. Outcomes from the study will help refine the design of a future definitive phase 3 trial. That future phase 3 trial will have a patient-centred primary endpoint, e.g. a meaningful improvement in Health Related Quality of Life (HRQOL) or an increase in treatment uptake or tolerance. Additional outcome measures are likely to include functional fitness, hospital admissions and overall survival.

A randomised prospective feasibility study will be performed over 12 months in two centres in the United Kingdom (Glasgow and Manchester). If eligible for the study, patients will be randomised 1:1 to receive a personalised exercise programme or standard care. Patients randomised to the intervention (exercise) arm will undergo an individualised assessment by either a physiotherapist or a qualified exercise specialist with specialised exercise and health condition qualifications. Following this initial assessment, patients will receive a tailored exercise, wellbeing and nutritional support package. The investigators will assess functional fitness and health-related quality of life scores as study outcome measures. The investigators also aim to conduct semi-structured interviews in patients who decline to participate or drop out of the study in order to examine barriers to study recruitment and retention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of mesothelioma, ratified by a mesothelioma multi-disciplinary team (MDT) meeting
2. Performance status 0 - 2
3. Clinical frailty score ≤5
4. Informed written consent

Exclusion Criteria:

1. Performance status ≥3
2. Clinical frailty score ≥6
3. Unlikely to be able to participate in an exercise programme (clinician/physiotherapist judgement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients recruited | 12 months
  Number of patients recruited to the study

SECONDARY OUTCOMES:
Proportion of screened patients who are ineligible | 12 months
  Proportion of screened patients who are ineligible for the study
Study drop-out rate | 12 months
  Proportion of patients who enter the study who withdraw prior to study completion
Intervention adherence rate | 12 months
  Proportion of patients randomised to the intervention arm who complete the exercise programme
Health-related Quality of Life questionnaire completion rate | 18 months
  Number of Health-related Quality of Life questionnaires completed by participants in the study (higher numbers of completed questionnaires equates to better outcome)
Framework analysis from qualitative interviews | 12 months
  Framework analysis from qualitative interviews with study participants

CONTACTS AND LOCATIONS:
Overall Officials: Selina Tsim, PhD, Principal Investigator — NHS Greater Glasgow & Clyde
Locations (2):
- United Kingdom (2):
  - Queen Elizabeth University Hospital, Glasgow
  - Wythenshawe Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nowak AK, Stockler MR, Byrne MJ. Assessing quality of life during chemotherapy for pleural mesothelioma: feasibility, validity, and results of using the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire and Lung Cancer Module. J Clin Oncol. 2004 Aug 1;22(15):3172-80. doi: 10.1200/JCO.2004.09.147. PMID 15284270
- [Background] Nagamatsu Y, Oze I, Aoe K, Hotta K, Kato K, Nakagawa J, Hara K, Kishimoto T, Fujimoto N. Quality of life of survivors of malignant pleural mesothelioma in Japan: a cross sectional study. BMC Cancer. 2018 Mar 27;18(1):350. doi: 10.1186/s12885-018-4293-x. PMID 29587685
- [Background] Hoon SN, Lawrie I, Qi C, Rahman N, Maskell N, Forbes K, Gerry S, Monterosso L, Chauhan A, Brims FJH. Symptom Burden and Unmet Needs in Malignant Pleural Mesothelioma: Exploratory Analyses From the RESPECT-Meso Study. J Palliat Care. 2021 Apr;36(2):113-120. doi: 10.1177/0825859720948975. Epub 2020 Aug 14. PMID 32791881
- [Background] Arnold DT, Hooper CE, Morley A, White P, Lyburn ID, Searle J, Darby M, Hall T, Hall D, Rahman NM, De Winton E, Clive A, Masani V, Dangoor A, Guglani S, Jankowska P, Lowndes SA, Harvey JE, Braybrooke JP, Maskell NA. The effect of chemotherapy on health-related quality of life in mesothelioma: results from the SWAMP trial. Br J Cancer. 2015 Mar 31;112(7):1183-9. doi: 10.1038/bjc.2015.77. PMID 25756395
- [Background] Baas P, Scherpereel A, Nowak AK, Fujimoto N, Peters S, Tsao AS, Mansfield AS, Popat S, Jahan T, Antonia S, Oulkhouir Y, Bautista Y, Cornelissen R, Greillier L, Grossi F, Kowalski D, Rodriguez-Cid J, Aanur P, Oukessou A, Baudelet C, Zalcman G. First-line nivolumab plus ipilimumab in unresectable malignant pleural mesothelioma (CheckMate 743): a multicentre, randomised, open-label, phase 3 trial. Lancet. 2021 Jan 30;397(10272):375-386. doi: 10.1016/S0140-6736(20)32714-8. Epub 2021 Jan 21. PMID 33485464
- [Background] Gravier FE, Smondack P, Prieur G, Medrinal C, Combret Y, Muir JF, Baste JM, Cuvelier A, Boujibar F, Bonnevie T. Effects of exercise training in people with non-small cell lung cancer before lung resection: a systematic review and meta-analysis. Thorax. 2022 May;77(5):486-496. doi: 10.1136/thoraxjnl-2021-217242. Epub 2021 Aug 24. PMID 34429375
- [Background] Olivier C, Grosbois JM, Cortot AB, Peres S, Heron C, Delourme J, Gierczynski M, Hoorelbeke A, Scherpereel A, Le Rouzic O. Real-life feasibility of home-based pulmonary rehabilitation in chemotherapy-treated patients with thoracic cancers: a pilot study. BMC Cancer. 2018 Feb 13;18(1):178. doi: 10.1186/s12885-018-4102-6. PMID 29433474
- [Background] Li S, Wang T, Tong G, Li X, You D, Cong M. Prognostic Impact of Sarcopenia on Clinical Outcomes in Malignancies Treated With Immune Checkpoint Inhibitors: A Systematic Review and Meta-Analysis. Front Oncol. 2021 Aug 26;11:726257. doi: 10.3389/fonc.2021.726257. eCollection 2021. PMID 34513704
- [Background] Jeffery E, Lee YCG, Newton RU, Lyons-Wall P, McVeigh J, Nowak AK, Cheah HM, Nguyen B, Fitzgerald DB, Creaney J, Straker L, Peddle-McIntyre CJ. Body composition and nutritional status in malignant pleural mesothelioma: implications for activity levels and quality of life. Eur J Clin Nutr. 2019 Oct;73(10):1412-1421. doi: 10.1038/s41430-019-0418-9. Epub 2019 Mar 18. PMID 30886321
- [Background] Mangano GD, Fouani M, D'Amico D, Di Felice V, Barone R. Cancer-Related Cachexia: The Vicious Circle between Inflammatory Cytokines, Skeletal Muscle, Lipid Metabolism and the Possible Role of Physical Training. Int J Mol Sci. 2022 Mar 10;23(6):3004. doi: 10.3390/ijms23063004. PMID 35328423
- [Background] Gerritsen JK, Vincent AJ. Exercise improves quality of life in patients with cancer: a systematic review and meta-analysis of randomised controlled trials. Br J Sports Med. 2016 Jul;50(13):796-803. doi: 10.1136/bjsports-2015-094787. Epub 2015 Dec 30. PMID 26719503
- [Background] Mishra SI, Scherer RW, Geigle PM, Berlanstein DR, Topaloglu O, Gotay CC, Snyder C. Exercise interventions on health-related quality of life for cancer survivors. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD007566. doi: 10.1002/14651858.CD007566.pub2. PMID 22895961
- [Background] Bradley P, Merchant Z, Rowlinson-Groves K, Taylor M, Moore J, Evison M. Feasibility and outcomes of a real-world regional lung cancer prehabilitation programme in the UK. Br J Anaesth. 2023 Jan;130(1):e47-e55. doi: 10.1016/j.bja.2022.05.034. Epub 2022 Jul 13. PMID 35840361
- [Background] Koller M, Musoro JZ, Tomaszewski K, Coens C, King MT, Sprangers MAG, Groenvold M, Cocks K, Velikova G, Flechtner HH, Bottomley A. Minimally important differences of EORTC QLQ-C30 scales in patients with lung cancer or malignant pleural mesothelioma - Interpretation guidance derived from two randomized EORTC trials. Lung Cancer. 2022 May;167:65-72. doi: 10.1016/j.lungcan.2022.03.018. Epub 2022 Mar 29. PMID 35413526

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT06491784/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT06491784/ICF_001.pdf